CLINICAL TRIAL: NCT02944331
Title: 3-4 Year Outcomes Following Endovenous Steam Ablation of the Saphenous Veins for the Treatment of Venous Insufficiency
Brief Title: 3-4 Year Outcomes Following Endovenous Steam Ablation for Venous Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Lovisenberg Diakonale Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Steam
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Varicose Veins
Keywords: Steam ablation; Endothermal ablation; Varicose vein treatment; Venous insufficiency; Saphenous vein reflux; Recurrent varicosity
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Endovenous steam ablation

SUMMARY:
The aim of this study is to evaluate the long-term effects of endovenous steam ablation (EVSA). Postoperative data at 3-4 year follow-up will be collected from patients treated with EVSA.

DETAILED DESCRIPTION:
Endovenous steam ablation (EVSA) of saphenous veins (saphenous vein reflux) is one of the endothermal methods in the modern treatment of venous insufficiency. Good results and long-term follow-up have been published for endovenous laser ablation (EVLA) and radiofrequency ablation (RFA), while long-term effects of EVSA are less documented. Therefore, the aim of this study is to evaluate the effect of EVSA in 200 consecutive patients treated with EVSA and conduct prospective evaluations at 3-4 year follow-up. Standardized and validated measures will be compared to preoperative measures to evaluate change in patient-reported and clinical outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

* Received steam ablation for treatment of saphenous vein reflux (clinical classes C2-C4) at Lovisenberg Diakonale Hospital 3-4 years (i.e, 36-48 months) prior to study enrollment.
* Ability to speak, understand, read, and write Norwegian in order to complete follow-up exams and questionnaires.

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received steam ablation for treatment of saphenous vein reflux (clinical classes C2-C4) 3-4 years prior to study enrollment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Vein obliteration or abolition of reflux | 3-4 years after treatment
  As determined by duplex scanning

SECONDARY OUTCOMES:
Recurrent varicosities | 3-4 years after treatment
Recanalization | 3-4 years after treatment
Venous Clinical Severity Score | 3-4 years after treatment
Aberdeen Varicose Vein Questionnaire | 3-4 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Lovisenberg Diakonale Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No